CLINICAL TRIAL: NCT06165055
Title: Investigation of Single Gene Polymorphisms Associated With Molar-Incisor Hypomineralization
Brief Title: Single Gene Polymorphisms Associated With Molar-Incisor Hypomineralization
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: MarmaraPedo2
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Molar-Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MIH-affected participants (study group ): The Study Arm comprises individuals aged 8-13 with Molar-Incisor Hypomineralization (MIH) in at least one permanent molar.
  Interventions: Diagnostic Test: DNA Sample Collection + DNA genotyping
- Systemically healthy controls (control group ): Systemically healthy individuals without MIH.
  Interventions: Diagnostic Test: DNA Sample Collection + DNA genotyping

INTERVENTIONS:
Diagnostic Test: DNA Sample Collection + DNA genotyping — Volunteers' oral epithelial cell DNA will be collected using DNA swabs, followed by DNA isolation with the PureLink DNA Isolation Kit. The isolated DNA's quality will be assessed using the Invitrogen QUBIT 4 Fluorometer, and the samples will be stored at -20°C until analysis of specific genetic regions.

SUMMARY:
The genetic factors associated with Molar-Incisor Hypomineralization (MIH), a dental condition affecting permanent molars in individuals aged 8-13. Buccal swab samples collected from 90 MIH-affected participants and 90 systemically healthy controls. The goal is to identify potential genetic markers contributing to the etiology of MIH, shedding light on previously unexplored aspects of genetic susceptibility.

DETAILED DESCRIPTION:
The aim of study is to elucidate the unknown aspects of genetic predisposition that may be effective in the etiology of Molar-Incisor Hypomineralization (MIH), that is, to identify unexplored genes that may be associated with MIH. The buccal swab method will be used for the purpose of collecting DNA samples.Samples will be collected from the inner cheek using a swab. The collected samples will be placed in single-use sterile Eppendorf tubes containing Phosphate Buffered Saline (PBS) solution. The samples will be stored at +4 degrees Celsius in a refrigerator, and DNA isolations will be performed within a few days. .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 8 and 13 years
* Patients whose parents consent to participate in the study
* Patients who provide cooperation for treatment and study
* For the study group: patients with at least one molar tooth showing molar-incisor hypomineralization
* For the control group: patients without molar-incisor hypomineralization
* Patients without a genetic disease in themselves or their family

Exclusion Criteria:

* Patients with a genetic disease in themselves or their family

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The Study Arm: healthy individuals aged 8-13 with Molar-Incisor Hypomineralization (MIH) in at least one permanent molar.
  The Control Arm: healthy individuals aged 8-13 without Molar-Incisor Hypomineralization (MIH).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
genotyping of polymorphisms | 1.5 -2 year
  The genotyping of polymorphisms will be conducted using the StepOnePlus instrument (Thermo Fisher Scientific, Inc.) through Real-Time PCR, following the manufacturers' protocols (cat. no. 4371355, Thermo Fisher Scientific, Inc.) and utilizing Taqman SNP genotyping kits. The reaction volume will be 10 µl in total, comprising 5 µl of Genotyping Master Mix (Applied Biosystems, Foster City, CA), 3.5 µl of nuclease-free H2O (Thermofisher, USA), 0.5 µl of genotyping assay (Applied Biosystems), and 1 µl of DNA.

IPD SHARING:
Plan to Share IPD: No